CLINICAL TRIAL: NCT02319824
Title: A Pilot Trial of NY-ESO-1-Specific T Cells in Patients With Metastatic NY-ESO-1-Expressing Sarcomas Receiving Palliative Radiation
Brief Title: NY-ESO-1-Specific T-cells in Treating Patients With Advanced NY-ESO-1-Expressing Sarcomas Receiving Palliative Radiation Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Seth Pollack, Responsible Party, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2721.00; NCI-2014-02154 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2721; 2721.00 (Other: Fred Hutch/University of Washington Cancer Consortium); K23CA175167 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2014-11-05; First posted 2014-12-18 (Estimated); Results first posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-04

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (radiation and NY-ESO-1-specific T cells) (Experimental): Patients undergo palliative radiation therapy at the discretion of the treating radiation oncologist. Patients then receive NY-ESO-1-specific T cells IV over 60 minutes 2-3 days after completion of radiation therapy.
  Interventions: Biological: Autologous NY-ESO-1-specific CD8-positive T Lymphocytes; Other: Laboratory Biomarker Analysis; Radiation: Palliative Radiation Therapy

INTERVENTIONS:
Biological: Autologous NY-ESO-1-specific CD8-positive T Lymphocytes — Given IV
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Palliative Radiation Therapy — Undergo palliative radiation therapy

SUMMARY:
This pilot, phase I trial studies the safety of cancer-testis antigen (NY-ESO-1)-specific T cells (a type of immune cell) in treating patients with NY-ESO-1-expressing sarcomas that have spread to other places in the body and are receiving palliative (relief of symptoms and suffering caused by cancer) radiation therapy. Placing a modified gene for NY-ESO-1 into white blood cells may help the body build an immune response to kill tumor cells that express NY-ESO-1. Palliative radiation therapy may help patients with advanced sarcoma live more comfortably. Giving NY-ESO-1-specific T cells following palliative radiation therapy may be a better treatment for patients with sarcomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and toxicity of NY-ESO-1-specific T cells when given following high-dose, hypo-fractionated palliative radiation to patients with advanced NY-ESO-1 expressing sarcomas.

SECONDARY OBJECTIVES:

I. To look for preliminary evidence of systemic efficacy of NY-ESO-1-specific T-cell therapy following radiation on non-radiated tumors.

II. To determine whether radiation increases trafficking of adoptively transferred NY-ESO-1-specific T cells by comparing tumor biopsy specimens from radiated and non-radiated tumors.

OUTLINE:

Patients undergo palliative radiation therapy at the discretion of the treating radiation oncologist. Patients then receive NY-ESO-1-specific T cells intravenously (IV) over 60 minutes 2-3 days after completion of radiation therapy.

After completion of study treatment, patients are followed up weekly for 2 weeks, at 4-6, 8, 10, and 12 weeks, and then for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA FOR SCREENING:

* Histopathological documentation of sarcoma
* Patients must express NY-ESO-1 in their tumor by immunohistochemistry (IHC) (> 5%) prior to leukapheresis
* For leukapheresis, patients must meet the following criteria (any exceptions to this will require prior approval by the apheresis director and principal investigator [PI]):
* Pulse > 45 or < 120
* Weight >= 45 kg
* Temperature =< 38° Celsius (C) (=< 100.4° Fahrenheit [F])
* White blood cell count (WBC) >= 2,000
* Hematocrit (HCT) >= 30%
* Platelets >= 75,000

INCLUSION CRITERIA FOR TREATMENT:

* A diagnosis of a metastatic or unresectable sarcoma
* Patient must have a biopsy-accessible tumor to be radiated
* Patient must have consulted with a radiation oncologist who is planning radiation; their radiation oncologist should have documented plans to administer a dose of at least 30 Gy in 5 or fewer fractions
* Human leukocyte antigen (HLA) type A0201 or A2402
* Zubrod (Eastern Cooperative Oncology Group [ECOG]) performance status of '0-2'
* All patients must have an electrocardiogram (ECG) within 2 weeks of starting conditioning
* All patients must have an echo or multigated acquisition (MUGA) scan showing ejection fraction (EF) > 50% and normal troponin and creatine kinase MB (CK MB) performed within 90 days of starting treatment

Exclusion Criteria:

EXCLUSION CRITERIA FOR SCREENING:

* Patients who do not meet the above inclusion criteria will not receive leukapheresis

EXCLUSION CRITERIA FOR TREATMENT:

* Patients with a history of proven myocarditis, pericarditis, or endocarditis
* Pregnant women, nursing women, men and women of reproductive ability who are unwilling to use effective contraception or abstinence; women of childbearing potential must have a negative pregnancy test within two weeks prior to study entry
* Inadequate renal function as indicated by serum creatinine >= 1.5 times the upper limit of normal
* Inadequate liver function as indicated by total bilirubin >= 1.5 times the upper limit of normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >= 2.5 times the upper limit of normal
* Active symptomatic congestive heart failure
* Clinically significant hypotension
* Newly diagnosed cardiac arrhythmia; patients with an arrhythmia that has been stable for at least 3 months will be allowed to participate
* Known untreated central nervous system (CNS) metastasis
* Patients with systemic infections requiring antibiotics or chronic maintenance/suppressive therapy
* Patients receiving systemic anticancer therapy (chemotherapy, "biologics", immunotherapy) less than 2 weeks prior to starting radiation
* Clinically significant autoimmune disorders requiring on-going systemic immune-suppression for control
* Patients with acquired immunodeficiency syndrome (AIDS) or who are known to be human immunodeficiency virus (HIV) positive are not eligible for this study; testing may have been done up to 3 months prior to treatment
* Current treatment with steroids
* Known infection with hepatitis B virus (HBV) and hepatitis C virus (HCV); testing may have been done up to 3 months prior to treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Pollack, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: NY-ESO-1 specific T cells
Groups:
- Treatment (Radiation and NY-ESO-1-specific T Cells): Patients undergo palliative radiation therapy at the discretion of the treating radiation oncologist. Patients then receive NY-ESO-1-specific T cells IV 2-3 days after completion of radiation therapy.
Period: Overall Study
Arm/Group | Treatment (Radiation and NY-ESO-1-specific T Cells)
Started | 2; 2 NY-ESO-1 specific T cells
Completed | 2; 2 NY-ESO-1 specific T cells
Not Completed | 0; 0 NY-ESO-1 specific T cells

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Radiation and NY-ESO-1-specific T Cells): Patients undergo palliative radiation therapy at the discretion of the treating radiation oncologist. Patients then receive NY-ESO-1-specific T cells 2-3 days after completion of radiation therapy.
  Autologous NY-ESO-1-specific CD8-positive T Lymphocytes
Arm/Group | Treatment (Radiation and NY-ESO-1-specific T Cells)
Number analyzed (Participants) | 2
Age, Customized [Mean (Full Range); unit: years] | 40 [27 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events Measured by the National Cancer Institute Common Terminology Criteria for Adverse Events Version (v)4.03
Description: CTCAE v4.03
Time Frame: Up to 12 weeks post-treatment
Population: treated patients
Measure: Number; unit: participants
Groups:
- Treatment (Radiation and NY-ESO-1-specific T Cells): Patients undergo palliative radiation therapy at the discretion of the treating radiation oncologist. Patients then receive NY-ESO-1-specific T cells I60 minutes 2-3 days after completion of radiation therapy.
Arm/Group | Treatment (Radiation and NY-ESO-1-specific T Cells)
Number analyzed (Participants) | 2
participants
  Grade 1 Rash (likely related) | 1
  Grade 2 Shortness of breath (possibly related) | 1
  Grade 2 Cough (possibly related) | 1
  Grade 1 Cough (probably related) | 1

2. Secondary Outcome: T Cell Transfer Based on Response Evaluation Criteria In Solid Tumors v1.1
Description: RECIST at 6 weeks after treatment (non-radiated tumors only)
Time Frame: At 6 weeks post-treatment
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Radiation and NY-ESO-1-specific T Cells): Patients undergo palliative radiation therapy at the discretion of the treating radiation oncologist. Patients then receive NY-ESO-1-specific T cells 2-3 days after completion of radiation therapy.
Arm/Group | Treatment (Radiation and NY-ESO-1-specific T Cells)
Number analyzed (Participants) | 2
Participants
  SD | 1
  PD | 1

3. Secondary Outcome: Transferred NY-ESO-1-specific T Cells Based on Flow Cytometry Using Major Histocompatibility Complex Tetramers
Description: Over 5% tet+ cells at 6 weeks? Patients may have detectable NY-ESO-1 specific T cells by MHC tetramers but if they are less than 5% this will be considered negative.
Time Frame: Up to 6 weeks post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Radiation and NY-ESO-1-specific T Cells)
Number analyzed (Participants) | 2
Participants
  Number of patients with <5% of CD8 T cells tet+ | 2
  >5% | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: CTCAE v4.03
Arm/Group | Treatment (Radiation and NY-ESO-1-specific T Cells)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Radiation and NY-ESO-1-specific T Cells) (N=2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) — 2 separate events in 1 patient, one grade 1 and one grade 2
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — grade 2

LIMITATIONS AND CAVEATS:
This trial was ended early as persistence was not at the level we had hoped and we had the opportunity to pursue a more promising strategy.

The data is limited by having only 2 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes